CLINICAL TRIAL: NCT05529927
Title: Efficacy and Safety of 24 Weeks Sustained-release Dexamphetamine in Patients With Moderate to Severe Cocaine Use Disorder With Comorbid Opioid Use Disorder - A Multicenter Randomized, Double-blind, Placebo-controlled Study
Brief Title: Efficacy and Safety of Sustained-release Dexamphetamine in Patients With Moderate to Severe Cocaine Use Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Parnassia Addiction Research Centre (Other)
Collaborators: Leiden University Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Radboud University Medical Center (Other); The Netherlands Cancer Institute (Other); Het Zwarte Gat (Unknown); Columbia University (Other)
Responsible Party: Principal Investigator, Peter Blanken, PhD, Senior researcher, Parnassia Addiction Research Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10140262110025
Record Dates: First submitted 2022-08-19; First posted 2022-09-07 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Cocaine Use Disorder
Keywords: cocaine use disorder; sustained-release dexamphetamine; agonist pharmacotherapy; opioid use disorder; methadone maintenance treatment; randomized controlled trial (RCT); placebo-controlled; double-blind
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sustained-release Dexamphetamine (Experimental): Tablets of 30 mg sustained-release dexamphetamine sulphate. Target dose: 90 mg/day, if tolerated. Tablets have to be taken daily, in the morning, per os for 24 weeks.
  Interventions: Drug: Sustained-release Dexamphetamine
- Placebo (Placebo Comparator): Identical matched placebo, dispensed under the same conditions and with similar frequency as the investigational product (see above).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sustained-release Dexamphetamine — During the first week, patients will be individually titrated to the target dose of 90 mg/day, if tolerated. From the second week onwards, patients are prescribed 3 tablets (30 mg) per day, if tolerated. Titration can be slower but should be finished at the end of week 4. After 4 weeks dosages can no longer be increased, and only be reduced.
  Patients will visit the treatment centre 2 times per week to take their study medication under supervision of the treatment staff and to receive take-home medication for the days in between study visits.
  After 24 weeks patients will be randomized to either (double-blind) continuation or discontinuation (placebo) of SR-Dexamphetamine treatment to assess the consequences of discontinuation, during a 6 weeks period.
  Arms: Sustained-release Dexamphetamine
Drug: Placebo — Dispensed under the same conditions and with similar frequency as the investigational product (see above).
  After 24 weeks study medication will be discontinued in the placebo group.
  Arms: Placebo

SUMMARY:
In The Netherlands, each year, about 15 thousand people come into treatment because of problems with cocaine use. There is no approved medication for treatment of cocaine addiction and the psychosocial treatment patients receive is not successful for everyone; many return to treatment several times. There is evidence that agonist ("replacement") medications are effective in treating addiction: methadone for heroin addiction; nicotine replacement for smokers. Dexamphetamine is a stimulant medication registered for treatment of ADHD. It may also be effective as agonist treatment for people with cocaine addiction.

It will be investigated whether sustained-release dexamphetamine in people with cocaine addiction, participating in routine methadone maintenance treatment for their comorbid opioid use disorder, (1) reduces cocaine use and (2) improves their health and quality of life.

DETAILED DESCRIPTION:
RESEARCH QUESTION/RATIONALE: Treatment for patients with cocaine use disorder is modestly effective and there is an urgent need for more effective treatments. Several randomized controlled trials, including our previous proof of principle study (Nuijten et al., 2016, The Lancet), suggest that sustained-release dexamphetamine is the most promising medication for the treatment of cocaine use disorder.

HYPOTHESIS & OBJECTIVES: Therefore, it is hypothesized that sustained-release dexamphetamine is effective in patients with cocaine use disorder in terms of reducing cocaine use and improving health and quality of life.

STUDY DESIGN: Multicentre randomized, double-blind, placebo-controlled study in 204 patients with cocaine use disorder - participating in routine methadone maintenance treatment for their comorbid opioid use disorder. In the 1st study phase (24 weeks) the efficacy and safety of sustained-release dexamphetamine is compared with placebo. In the 2nd double-blind, placebo-controlled randomized treatment discontinuation phase (6 weeks), we assess the consequences of discontinuation of sustained-release dexamphetamine treatment.

STUDY POPULATION: Patients with moderate/severe cocaine use disorder participating in routine oral methadone maintenance treatment for their comorbid opioid use disorder .

INTERVENTION: The investigational product is in tablets, containing 30 mg dexamphetamine sulphate in sustained-release formulation. Patients will be titrated to the target dose of 90 mg/day, if tolerated. Medication is dispensed twice weekly.

OUTCOME PARAMETERS: Primary endpoint: number of days of cocaine abstinence in the final 4 weeks of treatment, assessed by combined self-report and urinalysis. Key secondary endpoint: Good or improved overall health status (in terms of physical and mental health, and social functioning).

SAMPLE SIZE/DATA-ANALYSIS: Assuming 5 days difference in cocaine abstinent days in the final 4 weeks of the study to be clinically relevant requires 102 patients per treatment group in order to detect these 5 days difference (pooled standard deviation: 11 days; two-sided alpha=0.05; power=0.90). Primary analysis: The primary endpoint is modelled in a negative binomial regression analysis, with treatment group as independent variable and stratification variables (treatment centre, overall health status, and (nearly) daily cocaine use) as covariates.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients between 18 and 65 years of age;
* active participation in opioid agonist treatment with oral methadone;
* moderate or severe cocaine use disorder according to DSM-5;
* regular use of cocaine in the previous month (i.e., ≥8 days/month);
* snorting, inhaling or injecting cocaine use as primary route of administration;
* the intention to reduce or stop cocaine use;
* able and willing to attend the treatment centre for 2 days per week;
* able and willing to co-operate with the required study assessments and study procedures; and
* provide written informed consent.

Exclusion Criteria:

* severe medical (e.g., severe renal or kidney insufficiency/failure) or severe psychiatric problems (e.g. acute psychosis, current major depression, current bipolar disorder, acute suicidality);
* cardiovascular problems: clinically relevant ECG abnormalities, moderate to severe hypertension (SBP>140; DBP>90; HR>100), angina pectoris, history with myocardial infarction, CVA, heart failure;
* glaucoma;
* Gilles-de-la-Tourettesyndrome;
* pheochromocytoma;
* hyperthyroid status;
* current dyspnea;
* pregnancy or continued lactation;
* (indication for) treatment with other medications that might potentially be effective for stimulant use disorder (e.g., methylphenidate, disulfiram, bupropion, or modafinil);
* anticipated need for inpatient treatment (clinical judgement);
* (expected) inability to complete the 30 weeks study (e.g., due to expected incarceration or hospitalization);
* insufficient command of the Dutch language; and
* current participation in another addiction treatment study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
The number of days of cocaine abstinence | Final 4 weeks of treatment (first study phase; i.e., week 21-24)
  The number of days of cocaine abstinence in the final 4 weeks of treatment, assessed by combined self-report and urinalysis.

SECONDARY OUTCOMES:
Physical health | Final 4 weeks of treatment compared with baseline
  Physical health; self-reported, Maudsley Addiction Profile - Health Symptoms Scale (MAP-HSS)
Mental health | Final 4 weeks of treatment compared with baseline
  Mental health; self-reported, Brief Symptom Inventory (BSI)
Social functioning | Final 4 weeks of treatment compared with baseline
  Social functioning, criminality; self-reported, European Addiction Severity Index (EuropASI)

OTHER OUTCOMES:
Discontinuation: Proportion of patients with ≥5 days/month decrease in cocaine abstinent days | Final 4 weeks of treatment discontinuation phase (second study phase; i.e., week 27-30)
  Proportion of patients with ≥5 days/month decrease in cocaine abstinent days at end of discontinuation phase (compared with the number of cocaine abstinent days/month at the end of study phase 1; weeks 21-24).
Discontinuation: Proportion of patients in good or improved overall health status | Final 4 weeks of treatment discontinuation phase (second study phase; i.e., week 27-30)
  Proportion of patients in good or improved overall health status at end of discontinuation phase (compared with the proportion of patients in good or improved overall health at the end of study phase 1; weeks 21-24).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Blanken, PhD., Principal Investigator — Parnassia Addiction Research Centre

IPD SHARING:
Plan to Share IPD: Yes
Coded IPD will become available upon reasonable request. Procedures have not yet been determined.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Not yet determined.
Access Criteria: Not yet determined.

REFERENCES:
- [Background] Nuijten M, Blanken P, van de Wetering B, Nuijen B, van den Brink W, Hendriks VM. Sustained-release dexamfetamine in the treatment of chronic cocaine-dependent patients on heroin-assisted treatment: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 May 28;387(10034):2226-34. doi: 10.1016/S0140-6736(16)00205-1. Epub 2016 Mar 22. PMID 27015909
- [Background] Blanken P, Nuijten M, van den Brink W, Hendriks VM. Clinical effects beyond cocaine use of sustained-release dexamphetamine for the treatment of cocaine dependent patients with comorbid opioid dependence: secondary analysis of a double-blind, placebo-controlled randomized trial. Addiction. 2020 May;115(5):917-923. doi: 10.1111/add.14874. Epub 2020 Jan 6. PMID 31908066